CLINICAL TRIAL: NCT06812013
Title: Impact of Idiopathic Scoliosis on Balance and Footprint Symmetry in Adolescents
Status: Completed | Type: Observational
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Other Study IDs: Scoliosis
Record Dates: First submitted 2025-01-13; First posted 2025-02-06 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Scoliosis Idiopathic
Keywords: foot print; scoliosis; balance
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- healthy adolescents: healthy adolescents
  Interventions: Other: assessment of foot print and balance
- study group: adolescents with scoliosis
  Interventions: Other: assessment of foot print and balance

INTERVENTIONS:
Other: assessment of foot print and balance — For static and dynamic balance assessment, Biodex Medical Systems Inc., Shirley, New York, USA (serial n.: 13020193) was used. The device consists of a circular foot platform that permits tilting in all directions, height-adjustable support rails, height adjustable display screen, and a printer. Balance assessment by the Biodex system is a valid and reliable objective measurement.
  For assessment of foot print symmetry Tekscan HR walkway Mat™ pressure measurement system, Tekscan Inc. USA will be use. It is made up of a digital mat inserted into a wooden walkway, sensors (4 senses/cm2) embedded in the mat, and a computer running the Tekscan Software (version 7) for data extrapolation.

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is the most prevalent form of scoliosis that affects children after the age of 10 years and is considered a critical developmental stage of the musculoskeletal system of the child. AIS causes deviations in the CNS, leading to asymmetry of motor activity and, consequently, an incorrect position of the spine. The progressive deformation of the spine leads to increased asymmetry in body functions. This elevated asymmetry is understood by the nervous system as a norm, which causes children to cease to sense the correct body position that may affect both static and dynamic balance and the foot pressure symmetry of the child, which was not investigated in such cases in any previous studies till now.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic children and adolescents ages 10 to 18 years
* confirmed through X-rays; we focused on patients in growing age.
* adolescent idiopathic scoliosis that has a Cobb angle of 10° to 50°

Exclusion Criteria:

* Neuromuscular etiology (e.g., cerebral palsy, myelomeningocele, muscular dystrophy, spinal muscular atrophy, spina bifida, spinal cord injuries)
* Early-onset idiopathic etiology (infantile [ages 0 to 3 years] or juvenile [ages 4 to 9 years])
* Congenital etiology (e.g., hemivertebrae, failure of segmentation) Mesenchymal/syndromic etiology (e.g., Marfan syndrome, mucopolysaccharidosis, osteogenesis imperfecta, inflammatory diseases, postoperative)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population & Sample size: One hundred and fifty adolescents will be recruited to participate in the study, seventy-five of them will be healthy adolescents while the other Seventy-five adolescents will have idiopathic scoliosis with different degrees of scoliosis curves.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
static and dynamic balance | 2 months
  For static and dynamic balance assessment, Biodex Medical Systems Inc., Shirley, New York, USA (serial n.: 13020193) was used. The device consists of a circular foot platform that permits tilting in all directions, height-adjustable support rails, height adjustable display screen, and a printer. Balance assessment by the Biodex system is a valid and reliable objective measurement.
foot print | 2 months
  For assessment of foot print symmetry Tekscan HR walkway Mat™ pressure measurement system, Tekscan Inc. USA will be use. It is made up of a digital mat inserted into a wooden walkway, sensors (4 senses/cm2) embedded in the mat, and a computer running the Tekscan Software (version 7) for data extrapolation.

CONTACTS AND LOCATIONS:
Locations (1):
- Modern University for Technology and Information, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/books/NBK493371/table/appa.t8/